CLINICAL TRIAL: NCT07083947
Title: A Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Effect of Herbal Compositions CL19183 and CL24212 on Body Weight, Body Composition and Metabolic Health in Overweight Subjects
Brief Title: Effect of Herbal Compositions on Body Weight, Body Composition and Metabolic Health in Overweight Subjects
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ApexCPG LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: APX/OW/CL24212/25
Record Dates: First submitted 2025-07-11; First posted 2025-07-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): One capsule taken orally each morning after breakfast with water for 16 weeks
  Interventions: Other: Placebo
- CL19183 (Experimental): One capsule taken orally each morning after breakfast with water for 16 weeks
  Interventions: Dietary Supplement: CL19183
- CL24212 (Experimental): One capsule taken orally each morning after breakfast with water for 16 weeks
  Interventions: Dietary Supplement: CL24212

INTERVENTIONS:
Dietary Supplement: CL19183 — One capsule taken orally each morning after breakfast with water for 16 weeks
  Arms: CL19183
Dietary Supplement: CL24212 — One capsule taken orally each morning after breakfast with water for 16 weeks
  Arms: CL24212
Other: Placebo — One capsule taken orally each morning after breakfast with water for 16 weeks
  Arms: Placebo

SUMMARY:
The Purpose of the study is to evaluate the efficacy of herbal composition CL19183 and CL24212 on body weight, body composition and metabolic health in overweight subjects.

DETAILED DESCRIPTION:
A total of 150 male and female subjects aged between 25 and 55 years will be included in the study. Assessment of inclusion and exclusion criteria will be done based on clinical and laboratory investigations. The eligible subjects will be randomized as per the computer-generated randomization list. The subjects will be assigned to either CL19183:450 mg or CL24212:300 mg or Placebo arm at 1:1:1 ratio. The subjects will be instructed to take one capsule daily in the morning after breakfast for 16 weeks. Apart from primary and secondary outcomes, the study will also record the vital signs and adverse events to evaluate the herbal composition safety and tolerability. The safety assessment of the CL19183 and CL24212 will also include routine laboratory investigations on blood, urine and clinical chemistry at screening and the final visit of the intervention

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy male and female subjects aged between 25-55 years with body mass index (BMI) of 25-29.9 kg/m2.

  2. Subjects with sedentary lifestyle, no regular athletic or sports activities. 3. Subjects willing to participate in walking-exercise (5 days a week, 30 min per day) over study duration.

  4. Subjects with normal thyroid hormone profile. 5. Subjects agreed to consume recommended standard diet. 6. Subjects who are willing to abstain from alcohol, coffee, tea, cola, energy drinks & chocolate for at least 24 hrs. prior to visits and final visit.

  7. Subjects who are non-smokers. 8. Subject agrees to maintain diet tracker. 9. Subject considered generally healthy as per health history and routine clinical investigations during screening.

  10. Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, Depo-Provera®, or double-barrier and have a negative pregnancy test at the screening visit.

  11. Ability to understand the risks/benefits of the protocol and willing to sign the written informed consent.

Exclusion Criteria:

* 1. Subjects who were taking medications which affect the metabolic rate (e.g. antidepressants, beta-blockers, hormones, etc.).

  2. Subjects on weight loss practices, usage of weight reduction supplements/nutrition products will be excluded.

  3. Subjects underwent treatment for COVID 19 within last 3 months or tested positive during the study will be excluded.

  4. Subjects participated in any weight loss programs within 3 months. 5. Subjects who are diabetic and/or hypertensive. 6. Evidence or history of hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic diseases, malignancies.

  7. Subjects taking medications for or suffering from a medical condition that could impact results related to metabolism (e.g., thyroid disorders, diabetes, mental disorders such as anxiety or depression, heart disease, arthritis, cancer).

  8. Subjects with HIV Positive. 9. Female subjects, who are pregnant, breast feeding or planning to become pregnant during the study.

  10. Subjects having history of psychiatric disorder that may impair the ability of subjects to provide written informed consent.

  11. Any other condition that, in the opinion of the investigator, would adversely affect the subject's ability to complete the study or its measures.

  12. Use of nutritional supplements (e.g., creatine, protein drinks, amino acids, or vitamins) or ergogenic aids and caffeinated and not caffeinated thermogenics within 30 days prior to the study.

  13. Subjects who are participated or currently participating in another clinical trial within 30 days prior to screening.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to the end of the study period in Body weight | Week 0 (Baseline), Week 2, Week 4, Week 8, Week 12 & Week 16
  The subject's body weight is measured using a digital weighing scale. An improvement is indicated when the body weight falls within the normal range based on the subject's demographic characteristics.

SECONDARY OUTCOMES:
Change from baseline to the end of the study period in Body mass index (BMI) | Screening, Week 0 (Baseline),Week 2, Week 4, Week 8, Week 12 & Week 16
  Body mass index is a calculated measure by considering the weight and height of a subject. A change in BMI from overweight to normal range is a positive indicator of healthy lifestyle.
Change from baseline to the end of the study period in Body composition using DEXA (including fat and lean mass) | Week 0 (Baseline), Week 8& Week 16
  A low-dose X-ray is used to assess the fat and lean mass of a subject. An increase in lean mass indicates significant improvement, while a reduction in fat mass contributes to better overall health in the subject
Change from baseline to the end of the study period in Waist (WC) | Week 0 (Baseline),Week 2, Week 4,Week 8,Week 12,Week 16
  Waist circumference is measured around the abdomen, just above the navel. This value is influenced by the subject's height and weight. A reduction in waist circumference indicates improvement in body weight, as well as decreased fat storage and deposition.
Change from baseline to the end of the study period in Hip circumference (HC) | Week 0 (Baseline),Week 2, Week 4,Week 8,Week 12,Week 16
  It represents the maximum circumference measured around the buttocks. This measurement is influenced by the subject's height and weight. A reduction in this value indicates improvements in body weight, as well as a decrease in fat storage and deposition
Change from baseline to the end of the study period in Waist to hip ratio (WHR) | Week 0(Baseline), Week 2, Week 4, Week 8, Week 12& Week 16
  It's a ratio of waist to hip circumference. As the waist-to-hip ratio changes to the normal range according to person's demographic profile, this is associated with improvements in metabolism and body weight
Change from baseline to the end of the study period in Lipid profile (including amyloid A) | Week 0 (Baseline), Week 8 & Week 16
  Amyloid A (AA) is derived from serum amyloid A (SAA), an acute-phase reactant produced predominantly by the liver during inflammation, including obesity, which can lead to elevated levels of serum amyloid A (SAA). In AA amyloidosis, amyloid deposits typically affect the kidneys (leading to proteinuria and renal impairment.
Change from baseline to the end of the study period in Lipid profile (including Apo B) | Week 0 (Baseline), Week 8 & Week 16
  Apo B is a protein found on the surface of therogenic lipoproteins, including VLDL, IDL, LDL, and lipoprotein(a). It reflects the number of potentially harmful lipoprotein particles, making it a strong marker for cardiovascular risk due to obesity.
Change from baseline to the end of the study period in Adiponectin | Week 0 (Baseline), Week 8 & Week 16
  Adiponectin is a hormone secreted primarily by adipose (fat) tissue. It plays a crucial role in regulating glucose levels and fatty acid breakdown, contributing to metabolic health. Higher levels of adiponectin are associated with increased insulin sensitivity, anti-inflammatory effects, and reduced risk of cardiovascular disease
Change from baseline to the end of the study period in Ghrelin | Week 0 (Baseline), Week 8 & Week 16
  Ghrelin is a hormone primarily produced in the stomach, with smaller amounts secreted by other tissues such as the small intestine, pancreas, and brain. It is often referred to as the "hunger hormone" because it plays a key role in regulating appetite and energy balance. Abnormal ghrelin levels have been associated with conditions like obesity.
Change from baseline to the end of the study period in total glucagon-like peptide 1(GLP- 1) | Week 0 (Baseline), Week 8 & Week 16
  Glucagon-like peptide-1 (GLP-1) is an incretin hormone primarily produced in the intestinal L-cells in response to nutrient ingestion. It plays a significant role in glucose metabolism by stimulating insulin secretion, inhibiting glucagon release, slowing gastric emptying. GLP-1 influences weight management primarily by suppressing appetite, slowing gastric emptying, and reducing food intake.
Change from baseline to the end of the study period in C-Peptide | Week 0 (Baseline), Week 8 & Week 16
  C-peptide is a short chain of amino acids that is released into the bloodstream as a by-product when insulin is produced by the pancreas. During obesity, C-peptide levels are typically elevated due to increased insulin secretion driven by insulin resistance. Monitoring these levels can help assess β-cell function and the risk of progression to diabetes.
Change from baseline to the end of the study period in Glucagon | Week 0 (Baseline), Week 8 & Week 16
  Glucagon is a hormone produced by the alpha cells of the pancreas that primarily functions to increase blood glucose levels by stimulating hepatic glucose production. During weight loss, increased glucagon levels may be beneficial because It promotes the mobilization of stored fat by encouraging lipolysis.it helps maintain blood glucose levels when carbohydrate intake is reduced.
Change from baseline to the end of the study period in VCAM-1 | Week 0 (Baseline), Week 8 & Week 16
  VACM-1 is a cell surface glycoprotein expressed primarily on vascular endothelial cells in response to inflammatory stimuli. It plays a crucial role in mediating the adhesion and transmigration of leukocytes during inflammatory processes. In obesity, due to chronic low-grade inflammation, pro inflammatory cytokines such as IL-6, TNF-a induce the up regulation of adhesion molecules like VCAM-1 on endothelial cells lining blood vessels in adipose tissue.
Change from baseline to the end of the study period in ICAM- 1 | ICAM-1 is typically expressed at low levels on various cell types, including endothelial cells (lining blood vessels), immune cells (like leukocytes), and epithelial cells. ICAM-1 expression is significantly upregulated in adipose tissue in obesity.
  Day 1 (Baseline), Week 8 & Week 16

CONTACTS AND LOCATIONS:
Locations (1):
- Swaroop Rani Hospital, Motilal Nehru Medical College, Allahābād, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall KD, Guo J. Obesity Energetics: Body Weight Regulation and the Effects of Diet Composition. Gastroenterology. 2017 May;152(7):1718-1727.e3. doi: 10.1053/j.gastro.2017.01.052. Epub 2017 Feb 11. PMID 28193517
- [Background] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830
- [Background] Semlitsch T, Stigler FL, Jeitler K, Horvath K, Siebenhofer A. Management of overweight and obesity in primary care-A systematic overview of international evidence-based guidelines. Obes Rev. 2019 Sep;20(9):1218-1230. doi: 10.1111/obr.12889. Epub 2019 Jul 8. PMID 31286668